CLINICAL TRIAL: NCT03439111
Title: Standardized Lycium Chinense Fruit Extract Enhances Attention and Cognitive Function in Healthy Young People: A Double-blind, Randomized, Placebo-Controlled, Crossover Trial
Brief Title: Standardized Lycium Chinense Fruit Extract Enhances Attention and Cognitive Function in Healthy Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biomix (Industry)
Collaborators: Kyunghee University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KOMCGIRB-2013-88
Record Dates: First submitted 2018-02-01; First posted 2018-02-20 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Lycium chinense fruit
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Capsules

STUDY DESIGN:
Intervention Model Description: Participants receive one of two (or more) alternative interventions during the initial phase of the study and receive the other intervention during the second phase of the study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Intervention : Placebo + Standardized Lycium chinense Fruit Extract (LCF) capsules Placebo Comparator : Oral administration, 600 mg two capsules (600 mg of Starch/capsule) three times a day for 4 week treatment 3 week wash-out Experimental : Oral administration, 600 mg two capsules (146 mg of the Standardized Lycium chinense Fruit Extract (LCF)/capsule) three times a day for 4 week treatment
  Interventions: Dietary Supplement: Standardized Lycium chinense Fruit Extract (LCF) capsules
- Experimental (Experimental): Intervention : Standardized Lycium chinense Fruit Extract (LCF) capsules + Placebo Experimental : Oral administration, 600 mg two capsules (146 mg of the Standardized Lycium chinense Fruit Extract (LCF)/capsule) three times a day for 4 week treatment 3 week wash-out Placebo Comparator : Oral administration, 600 mg two capsules (600 mg of Starch/capsule) three times a day for 4 week treatment
  Interventions: Dietary Supplement: Standardized Lycium chinense Fruit Extract (LCF) capsules

INTERVENTIONS:
Dietary Supplement: Standardized Lycium chinense Fruit Extract (LCF) capsules — All dried water extracts and capsules of the Standardized Lycium chinense Fruit Extract (LCF) and Standardized Lycium chinense Fruit Extract (LCF)-matched placebo capsules used in the present study were manufactured and provided by the BIOMIX Company (Ilsan City, Korea).

SUMMARY:
Lycium chinense fruit (LCF) is widely distributed in East Asia that has been used traditionally for anti-aging purposes. This study was performed to examine the effects of LCF on attention and cognitive function in healthy young people. An 11-week, double-blind, randomized, placebo-controlled, crossover trial was conducted.

DETAILED DESCRIPTION:
The Computerized Neurocognitive function Test (CNT), the Korean version of the Attention-deficit/hyperactivity disorder (ADHD) Rating Scale-IV (K-ADHD-RS-IV), the Clinical Global Impression (CGI) rating scale, the Frankfurt Attention Inventory (FAIR), and resting-state electroencephalogram (EEG) were conducted before and after the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 14 and 24 years old
* Male or female
* Ability to understand the objectives of the study and agreed to abide by the required rules during the study.
* If participants were aged between 14 and 20 years old, they and their parents had to provide informed consent.

Exclusion Criteria:

* Diagnosis of ADHD (any subtype) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria
* Diagnosis of a developmental disorder
* Pregnant or breastfeeding women and women with the possibility of getting pregnant
* Gastrointestinal disease or history of gastrointestinal surgery, which might affect the absorption of study materials
* Significant neurological (epilepsy, mental retardation, or stroke) or medical illnesses (diabetes, hypertension, or cardiovascular diseases),
* Participation in other clinical studies during the four weeks preceding the start of the study
* More than 1.5 times normal limit of ALT or AST.

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2013-04-30 (Actual); Study Completion 2013-04-30 (Actual)

PRIMARY OUTCOMES:
The Computerized neurocognitive Function Test (CNT) | Before treatment, 4 and 11 weeks after treatment
  Change of its total score or its subscale score before treatment, 4 and 11 weeks after treatment

SECONDARY OUTCOMES:
Korean version of Attention-deficit/hyperactivity disorder (ADHD) Rating Scale-IV (K-ADHD-RS-IV) | Before treatment, 4 and 11 weeks after treatment
  Change of its total score or its subscale score before treatment, 4 and 11 weeks after treatment
The Clinical Global Impression (CGI) rating scale | Before treatment, 4 and 11 weeks after treatment
  Change of its total score or its subscale score before treatment, 4 and 11 weeks after treatment
The Frankfurt Attention Inventory (FAIR) | Before treatment, 4 and 11 weeks after treatment
  Change of its total score or its subscale score before treatment, 4 and 11 weeks after treatment
Resting-state electroencephalogram (EEG) | Before treatment, 4 and 11 weeks after treatment
  Change of its total score or its subscale score before treatment, 4 and 11 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hun Cho, KMD., Ph.D., Principal Investigator — Kyunghee University
Locations (1):
- Biomix, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No